CLINICAL TRIAL: NCT07308067
Title: Kinetics of Transmural Healing in Patients With Crohns Disease Treated With Risankizumab (SKYRIZI®)
Acronym: SKYNETICS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2025 BUISSON_CF533
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Crohn Disease (CD); Transmural Response
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Crohn's disease (CD) is a chronic inflammatory bowel disease (IBD) that can highly alter patients' quality of life and lead to bowel damage due to its transmural pattern. The current guidelines recommend to use treat-to-target strategies to achieve the combination of steroid-free clinical remission and endoscopic remission. However, the implementation of these strategies and endpoints are limited by the need of repeated colonoscopies, which dramatically reduced patients' acceptability and adherence to such a management. The concept of transmural healing has emerged as a promising therapeutic target. It has been associated with longer time spent in steroid-free clinical remission, decreased risk of hospitalization, slower progression of bowel damage and reduced risk of subsequent surgery. Furthermore, recent works suggested that transmural healing could lead to better outcomes, such as prevention of bowel damage progression, than endoscopic remission. Recently, the DEVISE-CD project proposed validated definitions of transmural healing and response (TR50 and TR25) using the modified Clermont score (C-score). Thus, transmural healing will become the next reference target in the near future. Although most data were generated using MRI, intestinal ultrasound (IUS) is an interesting alternative to assess transmural response thanks to its lower cost and high patients' acceptability enabling repeated procedures. IUS is now part of routine practice in day-care units.

Recently, Risankizumab, the first in-class anti-IL23 targeting p19 subunit in CD, demonstrated high level of efficacy to achieve and maintain clinical and endoscopic remission. However, no data are hitherto available on the kinetics and the efficacy of risankizumab to achieve transmural healing.

DETAILED DESCRIPTION:
This will be a prospective, multicenter study (5 centers) based on routine clinical practice, without any additional procedures. Data will be collected from electronic medical records and entered in a pseudonymized manner into the electronic case report form (RedCAP).

The data collected in this study include: demographic data (age, sex); disease-related data (date of diagnosis, disease duration, location, and phenotype); data on risankizumab treatment (start date, dosage, adverse events); clinical data (symptoms); laboratory data (CRP and fecal calprotectin); and radiological data (intestinal ultrasounds). These data will be collected, when available, at treatment initiation with SKYRIZI, and at weeks 4 and 12 as part of routine care.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients (≥ 18 years old) diagnosed with Crohns disease according to ECCO guidelines
* Initiating risankizumab therapy in routine practice
* Undergoing IUS procedures before and after risankizumab therapy

Exclusion Criteria:

* Ulcerative colitis and unclassified colitis
* Follow-up shorter than 3 months (except for those discontinuing risankizumab due to side effect or failure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Crohn's disease initiating treatment with risankizumab.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Transmural response evaluated by IUS at week 4 and 12. | From enrollment to the end of induction at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Buisson, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (4):
- France (4):
  - Amiens university hospital, Amiens
  - Clermont-Ferrand University hospital, Clermont-Ferrand
  - Grenoble university hospital, Grenoble
  - Marseille University Hospital, Marseille